CLINICAL TRIAL: NCT05528016
Title: Elaborated Analysis of Short and Long-term Results of Skin Versus Skin Plus Orbicularis Resection Blepharoplasty on Corneal Nerves, Meibomian Glands, Dry Eye Parameters, and Eyebrow Position
Brief Title: Short and Long-term Results of Skin Versus Skin Plus Orbicularis Resection Blepharoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09.2022.102
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Dermatochalasis of Eyelid; Ocular Surface Disease; Meibomian Gland Dysfunction; Dry Eye; Brow Ptosis
Keywords: blepharoplasty; skin; orbicularis oculi; corneal confocal microscopy; meibomian gland; dry eye; eyebrow
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Masking Description: All evaluations and data collection were performed by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin-Only Blepharoplasty (Active Comparator): Only the skin excision was performed for upper eyelid dermatochalasis.
  Interventions: Procedure: Upper Eyelid Blepharoplasty
- Skin+Muscle Blepharoplasty (Active Comparator): Skin plus muscle excision was performed for upper eyelid dermatochalasis.
  Interventions: Procedure: Upper Eyelid Blepharoplasty

INTERVENTIONS:
Procedure: Upper Eyelid Blepharoplasty — Blepharoplasty is a procedure that the skin, orbicularis oculi muscle, and fat pads are excised to treat visual field loss caused by dermatochalasis.

SUMMARY:
This study aims to evaluate the short and long-term effects of skin-only and skin+muscle excision blepharoplasty on corneal nerves, dry eye parameters, meibomian glands, and eyebrow position.

DETAILED DESCRIPTION:
The study was designed with the approval of the Ethics Committee on Human Research of Marmara University and was conducted following the tenets of the Declaration of Helsinki. Written informed consent was obtained from all patients who received information about the procedure and the postoperative course. The study included 48 eyes of 24 patients older than 18 who applied to Marmara University Oculoplastic and Orbital Surgery Unit due to dermatochalasis and were suggested upper eyelid blepharoplasty for medical or cosmetic purposes. The patients were divided into two groups, Group S (n=12) for skin excision only and Group M (n=12) for skin+muscle excision by the decision of the surgeon. In addition to all ophthalmological examinations, sub-basal nerve plexus parameters with corneal confocal microscopy, Schirmer I test, non-invasive tear break-up time, meibomian gland area loss measurements with infrared meibography, central eyebrow height, and lateral eyebrow height were evaluated at baseline and postoperative 1st week, 1st month and 1st-year follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18.
* Patients with dermatochalasis.
* Patients who were suggested upper eyelid blepharoplasty for medical or cosmetic purposes.

Exclusion Criteria:

* Patients who have had previous periorbital or ophthalmic surgery
* Patients with extensive blepharitis
* History of contact lens use
* History of ophthalmic, endocrinological, neurological, or rheumatological diseases
* History of facial paralysis
* Negative Bell's phenomenon
* Schirmer test <5mm
* The patients who had been treated with periocular botulinum toxin in the last 1 year were not included the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Corneal nerve fiber density (CNFD) | Baseline / 1 Week / 1 Month / 1 Year
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; University of Manchester, Manchester, UK) was used to analyze CNFD in fibers/mm2
Corneal nerve branch density (CNBD) | Baseline / 1 Week / 1 Month / 1 Year
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; University of Manchester, Manchester, UK) was used to analyze CNBD in branches/mm2.
Corneal nerve fiber length (CNFL) | Baseline / 1 Week / 1 Month / 1 Year
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; University of Manchester, Manchester, UK) was used to analyze CNBD in mm/mm2.
Eyebrow position | Baseline / 1 Week / 1 Month / 1 Year
  Millimetric measurement was performed to evaluate the effect of blepharoplasty on eyebrow position.
Meibomian Gland Area Loss (MGAL) | Baseline / 1 Week / 1 Month / 1 Year
  Phoenix-Meibography Imaging software that is available in the Sirius® Scheimpflug topographer (Sirius, CSO, Italy) was used to evaluate meibomian gland area loss in percentage.
Non-invasive Tear Break-Up Time (NI-BUT) | Baseline / 1 Week / 1 Month / 1 Year
  Phoenix-Meibography Imaging software that is available in the Sirius® Scheimpflug topographer (Sirius, CSO, Italy) was used to evaluate non-invasive tear break-up time in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Dericioğlu, M.D, Principal Investigator — Marmara University
Locations (1):
- Marmara University Pendik Research and Educational Hospital, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data supporting the study findings are available from the corresponding author upon request.

REFERENCES:
- [Derived] Dericioglu V, San B, Sevik MO, Akkaya Turhan S. Skin-Only Versus Skin-Plus-Orbicularis Resection Blepharoplasty: An Elaborated Analysis of Early- and Long-Term Effects on Corneal Nerves, Meibomian Glands, Dry Eye Parameters, and Eyebrow Position. Ophthalmic Plast Reconstr Surg. 2023 Sep-Oct 01;39(5):479-486. doi: 10.1097/IOP.0000000000002376. Epub 2023 Mar 27. PMID 36972140